CLINICAL TRIAL: NCT00697528
Title: Color Doppler Imaging of Orbital Venous Flow in Grave's Orbitopathy
Status: Completed | Type: Observational
Sponsor: University of Sao Paulo (Other)
Responsible Party: Hélio Angotti Neto, HCFMUSP - University of São Paulo
Other Study IDs: 352/06
Record Dates: First submitted 2008-06-11; First posted 2008-06-16 (Estimated); Last update posted 2013-12-19 (Estimated); Status verified 2008-06

CONDITIONS: Graves' Disease; Graves' Ophthalmopathy
Keywords: Graves; Color Doppler Imaging; Graves' Ophthalmopathy; Orbital Venous Flow
MeSH Terms: conditions — Graves Disease; Graves Ophthalmopathy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Group control with healthy subjects: Healthy subjects without thyroid disease, ocular disease and previous surgery in the orbit or eye used in the study.
- Graves' Ophthalmopathy - fibrotic phase: Patients that are clinically inactive (CAS equal or lower than 2). This group will be subdivided in the miogenic and lipogenic groups.
- Graves' Ophthalmopathy - active phase: Patients that are clinically active, presenting a CAS of 4 or more points, with or without disthyroid optic neuropathy.

SUMMARY:
Orbital Venous flow study in patients with Grave's Orbitopathy in different manifestation forms and stages, made with Color Doppler Imaging

DETAILED DESCRIPTION:
Prospective study with Grave's patients in active and fibrotic disease, myogenic and lipogenic forms, with muscle restriction and without muscle restriction and with or without optic compressive neuropathy. Blood flow was studied with Color Doppler Imaging (CDI) in the following orbital vessels:

* Superior Ophthalmic Vein (main target of the study protocol)
* Retinal Central Vein
* Retinal Central Artery
* Ophthalmic Artery

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Grave's Orbitopathy with well defined disease.

Exclusion Criteria:

* Uncertain cases, with an undefined status of Grave's Ophthalmopathy.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with Grave's disease within the orbital service of HCFMUSP at the Ophthalmology Department
Sampling Method: Non-Probability Sample
Enrollment: 66 (Actual)
Dates: Start 2007-01; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mário LR Monteiro, Professor, Study Director — Instituto do Coracao; Joseph E Benabou, Study Chair — Instituto do Coracao
Locations (1):
- Hospital das Clínicas da Universidade São Paulo, São Paulo, São Paulo, Brazil

REFERENCES:
- [Derived] Monteiro ML, Moritz RB, Angotti Neto H, Benabou JE. Color Doppler imaging of the superior ophthalmic vein in patients with Graves' orbitopathy before and after treatment of congestive disease. Clinics (Sao Paulo). 2011;66(8):1329-34. doi: 10.1590/s1807-59322011000800004. PMID 21915479